CLINICAL TRIAL: NCT01093391
Title: A Randomized Trial of Bare Metal Stent (Cronus®) - Cobalt Chromium Versus Stent Coating With Sirolimus (DES)
Brief Title: A Trial of Bare Metal Stent - Cobalt Chromium Versus Stent Coating With Sirolimus
Acronym: INSPIRON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Scitech 001
Record Dates: First submitted 2010-03-18; First posted 2010-03-25 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery; thrombosis; stent
MeSH Terms: conditions — Coronary Artery Disease; Thrombosis | interventions — Drug-Eluting Stents; Angiography; Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BARE METAL STENT (Placebo Comparator): BARE METAL STENT - STENT CRONUS
  Interventions: Device: BARE METAL STENT
- DRUG ELUTING STENT (Experimental): STENT INSPIRON WITH SIROLIMUS
  Interventions: Device: DRUG ELUTING STENT

INTERVENTIONS:
Device: DRUG ELUTING STENT — Site preparation and percutaneous access should be performed as per standard hospital procedures.It is recommended to cross the target lesion with 0.014-inch exchange-length guide wire. The involved lesion should be predilated with appropriately sized balloons using standard techniques. It is strongly encouraged that the Investigators use similar materials and techniques throughout the study to maintain consistency and standardization of care.A stent consists of an endovascular prosthesis with a metallic mesh structure that is implanted at the site of the artery blockage via catheterization procedure. The objective of stenting is to obtain an angiographic appearance of the expanded stent only outside the limits of the target vessel filled with contrast medium.
  Other Names: Angiography, Stenting
  Arms: DRUG ELUTING STENT
Device: BARE METAL STENT — Site preparation and percutaneous access should be performed as per standard hospital procedures.It is recommended to cross the target lesion with 0.014-inch exchange-length guide wire. The involved lesion should be predilated with appropriately sized balloons using standard techniques. It is strongly encouraged that the Investigators use similar materials and techniques throughout the study to maintain consistency and standardization of care.A stent consists of an endovascular prosthesis with a metallic mesh structure that is implanted at the site of the artery blockage via catheterization procedure. The objective of stenting is to obtain an angiographic appearance of the expanded stent only outside the limits of the target vessel filled with contrast medium.
  Arms: BARE METAL STENT

SUMMARY:
The objective of this study is to evaluate the security issues and efficacy of coronary stenting Cobalt Chrome covered with sirolimus-eluting Cobalt Chrome platform in patients with coronary artery lesion.

DETAILED DESCRIPTION:
Patients will be treated in compliance with the eligibility criteria, with stent study of 16-19mm. All patients are clinically followed for 60 months after the procedure and will undergo a control angiography 6 months. Can be treated multiple lesions, measuring between 2.5-3.5mm (by visual estimate). Patients enrolled will be randomized in a 1:2 propose in one of the groups with or without stent coating, respectively. And a randomized clinical trial, prospective study in 5 centers including 60 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤75 years;
2. Symptomatic cardiac ischemic disease and/or documented evidence of myocardial ischemia;
3. Types B1 and B2 coronary lesions (according to the ACC/AHA classification modified by Ellis);
4. Target lesion located in a native coronary artery;
5. Target lesion in vessel with diameter ranging from 2.5 to 3.5 mm (by visual estimate) amenable to treatment (coverage) with a 16- 19mm-long stent;
6. Target lesion with >50% diameter stenosis (by visual estimate);
7. Acceptable candidate to myocardial revascularization surgery (coronary artery bypass graft surgery);
8. The subject has been fully informed of the nature of the study, is willing to comply with all study requirements and will provide written informed consent as approved by the Ethics Committee of the respective clinical site.

Exclusion Criteria:

1. Female patients of childbearing potential;
2. Recent Q-wave myocardial infarction occurred within 48 hours prior to the index procedure. Recent Q-wave or non-Q-wave myocardial infarction with still elevated levels of cardiac markers;
3. Documented left ventricular ejection fraction <30%;
4. Renal dysfunction (creatinine > 2.0 mg/dL or 177 µmol/L);
5. Platelet count <100,000 cells/mm³ or >700,000 cells/mm³.;
6. White blood cell count <3,000 cells/mm3;
7. Suspected or documented hepatic disease (including laboratorial evidence of hepatitis);
8. Heart transplant receptor;
9. Known hypersensitivity to cobalt-chromium or to medications such as aspirin, clopidogrel bisulfate (Plavix or ISCOVER), ticlopidine (Ticlid) or heparin.
10. Concurrent medical condition with a life expectancy of less than 12 months;
11. Any major medical condition that, in the Investigator's opinion, may interfere with the optimal participation of the patient in this study;
12. Subject is currently participating in an investigational drug or another device study, including planned participation in an investigational drug or another device study during the course of the present investigation;
13. Coronary angioplasty (with or without stenting) less than 9 months before the index procedure at any site of the target vessel;
14. Previous coronary angioplasty (with or without stenting) at any time (>9 months) in a vessel segment less than 5 mm proximal or distal to the target lesion.
15. Planned coronary angioplasty (with or without stenting) in the first 12 months after the index procedure in any segment of the target vessel;

4.3. ANGIOGRAPHIC EXCLUSION CRITERIA

1. Restenotic target lesion;
2. More than one lesion requiring treatment in the same vessel;
3. Target vessel diameter <2.5 mm or >3.5 mm (by visual estimation);
4. Long target lesion not amenable to treatment (coverage) with a 16-19mm long stent;
5. Unprotected coronary artery branch lesion (≥50% diameter stenosis)
6. Target lesion is located in a surgical bypass graft;
7. Total vessel occlusion (TIMI flow grade 0-1);
8. Target lesion with ostial location;
9. Target lesion located in a lateral branch bifurcation >2.5mm or requiring lateral branch stenting;
10. Calcified target lesion that anticipates unsuccessful/impracticable predilation;
11. Target vessel with excessive tortuosity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Lumen Loss | 6 months after the procedure
  For an accurate assessment of the stent conditions 6 months after implantation, a follow-up catheterization will be performed at the 6-month visit in order to measure the diameter of the artery at the stented site. The objective is the lumen loss in-segment (including the portion in-stent and edges of 5 mm proximal and distal) at 6 months.

SECONDARY OUTCOMES:
Adverse Cardiac Events | 30 days, 6, 12 and 60 months after the procedure
  The clinical follow-up should be performed during the index procedure at 30 days, 6, 12 and 60 months post-procedure, and should consist of an assessment of the angina status (according to the Canadian Cardiovascular Society Classification and the Braunwald Classification for unstable angina) and major adverse cardiac events and any interventional treatment (e.g.: repeated target lesion revascularization or recurrent ischemia).

CONTACTS AND LOCATIONS:
Overall Officials: Expedito E. Ribeiro da Silva, Medicine, Principal Investigator — Instituto do Coração do Hospital das Clínicas da Fac. de Medicina da USP
Locations (4):
- Brazil (4):
  - Hospital Ibiapaba de Barbacena, Barbacena, Minas Gerais
  - Instituto de Assistêcia Médica ao Servidor Publico Estadual, São Paulo, São Paulo
  - Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo

REFERENCES:
- [Result] Carlos Augusto Homem de Magalhães Campos; Celso K. Takimura; Guilherme B. Gregores; Carlos A. Sarmento; Emerson T. Fioretto; Fracisco R. M. Laurindo; Expedito E. Ribeiro; Eulógio E. Martinez; Thiago F.C.C. Borges; Pedro A. Lemos. Redução neointimal com Stent com polímero biodegradável e Sirolimus desenvolvido no Brasil: Resultados preliminares em Suínos. Rev. Soc. Cardiol. Estado de São Paulo - Supl. B - Vol. 19
- [Derived] Oliveira MD, Ribeiro EE, Campos CM, Ribeiro HB, Faillace BL, Lopes AC, Esper RB, Meirelles GX, Perin MA, Abizaid A, Lemos PA. Four-year clinical follow-up of the first-in-man randomized comparison of a novel sirolimus eluting stent with abluminal biodegradable polymer and ultra-thin strut cobalt-chromium alloy: the INSPIRON-I trial. Cardiovasc Diagn Ther. 2015 Aug;5(4):264-70. doi: 10.3978/j.issn.2223-3652.2015.07.05. PMID 26331110
- [Derived] Ribeiro EE, Campos CM, Ribeiro HB, Lopes AC, Esper RB, Meirelles GX, Perin MA, Abizaid A, Lemos PA. First-in-man randomised comparison of a novel sirolimus-eluting stent with abluminal biodegradable polymer and thin-strut cobalt-chromium alloy: INSPIRON-I trial. EuroIntervention. 2014;9(12):1380-4. doi: 10.4244/EIJV9I12A234. PMID 24755382
- See also: Sponsor site — http://www.scitechmed.com
- See also: Site about the location that will be done the study. Location where the principal investigator works. — http://www.incor.usp.br
- See also: National Information System on Ethics in Research involving Human — http://portal2.saude.gov.br/sisnep/